CLINICAL TRIAL: NCT03552198
Title: Improving the Behavioural Impact of Air Quality Alerts in London
Brief Title: Improving the Behavioural Impact of Air Quality Alerts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: LRS-16/17-4286
Record Dates: First submitted 2018-05-15; First posted 2018-06-11 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2018-05

CONDITIONS: Pollution; Exposure; Health Behavior
Keywords: Air quality alerts; Health behaviour change; Adherence
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: This was a randomised control trail using a 2-way factorial design, with target population (2 levels: general population vs. individuals with a pre-existing health condition) and message format (2 levels: usual message format vs. alternative format) as between-factors.
Who Masked: Participant
Masking Description: To avoid bias participants were not told how the wording of the health advice had been changed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- General public/usual health advice (No Intervention): Healthy participants with a self-reported existing health condition were randomised to receive the usual UK Air Quality Indices health advice.
- General public/alternative health advice (Experimental): Generally healthy participants were randomised to receive targeted health advice about the adoption of protective behaviours in an alternative format.
  Interventions: Behavioral: Alternative health advice
- At risk group/usual health advice (No Intervention): Participants with a self-reported pre-existing health condition were randomised to receive the usual UK Air Quality Indices health advice.
- At risk group/alternative health advice (Experimental): Participants with a self-reported existing health conditions were randomised to receive targeted health advice (based on their health condition) about the adoption of protective behaviours in an alternative format.
  Interventions: Behavioral: Alternative health advice

INTERVENTIONS:
Behavioral: Alternative health advice — These messages targeted specific beliefs about air pollution and protective actions aimed at reducing exposure to air pollution. In addition, message specificity was targeted, which means that compared to the usual messages, the alternative messages reported more detailed health recommendations.
  Arms: At risk group/alternative health advice; General public/alternative health advice

SUMMARY:
The evidence shows that adherence to air quality advice to adopt protective behaviours during pollution episodes is suboptimal, and that the traditional strategy of simply informing people about high pollution episodes is not effective. The aim of the present study was to investigate how to improve the behavioural impact of existing air quality alert messages through a systematic manipulation of key communication variables, including perceived susceptibility, self-efficacy, response efficacy, planning, message specificity, etc. Users of an existing air quality alert smartphone application in London, who agreed to take part in the study, were randomly allocated to a control group (i.e. receiving usual health advice associated with the official UK Air Quality Index) or an intervention group receiving health advice associated with air quality alerts in an alternative format (i.e. targeting key variables). Both intended and actual adherence behaviours were investigated. Qualitative data were also collected to understand the reasons for not adopting protective behaviours in response to receiving a real air pollution alert.

Implications of this study include the potential to increase protective behaviours in the general population during air pollution episodes through the development of more effective communication strategies provided via existent air quality alert systems.

DETAILED DESCRIPTION:
According to data released in 2014, in 2012 around 3.7 million people died prematurely in the world as a result of exposure to ambient air pollution ((WHO), 2014). Evidence has shown the negative short- and long-term effects of air pollution on both premature mortality and morbidity from cardiopulmonary disease (for an overview, see (Kelly & Fussell, 2015)). This is particularly a problem in London (Samoli et al., 2016), where levels of air pollution are quite worrying. In the UK monitoring networks measure the levels of different air pollutants, and these measurements are provided by the Department for Environment, Food & Rural Affairs (DEFRA) in the form of daily air quality indices (AQIs), together with separate health advice for at-risk groups and the general population. A recently published systematic review (D'Antoni, Smith, Auyeung, & Weinman, 2017) has found suboptimal adherence levels to health advice associated with air quality alerts, and identified several facilitators and barriers of adherence. Some of the facilitators included beliefs that air pollution can have negative health effects (i.e. perceived severity), outcome expectancies (e.g., beliefs that something can be done to reduce smog), beliefs about the health benefits of AQI adoption (i.e. response efficacy), and receiving advice from health care professionals. Barriers to adherence included: lack of understanding of the indices, being exposed to health messages that reduced both concern about air pollution and perceived susceptibility, as well as perceived lack of self-efficacy/locus of control, reliance on sensory cues and lack of time to make behavioural changes. The findings of this systematic review have informed the current research study, which aimed to improve the behavioural impact of existing air quality alerts. In particular, alternative health messages were developed based on the psychosocial factors identified in the systematic review. The purpose of the study was to test whether these theory and evidence-based alternative communication formats, compared to the official messages sent in association with the UK AQIs, maximise the behavioural impact of existing alert systems.

Methods

Design:

This was a randomised control trail using a 2-way factorial design, with target population (2 levels: general population vs. individuals with a pre-existing health condition) and message format (2 levels: usual message format vs. alternative format) as between-factors. Qualitative data were also collected to understand the reasons for actual adherence and non-adherence.

- Theoretical framework and targeted psychosocial predictors:

The COM-B model (Michie, van Stralen, & West, 2011) was used as a theoretical framework to guide in the understanding of the facilitators and barriers to behaviour change in response to air quality alerts. The control groups received usual air quality alerts and health advice based on the UK AQI messages, and the intervention groups received alternative health messages targeting knowledge about the health impact of exposure to air pollution, perceived severity of air pollution, perceived susceptibility, perceived efficacy of protective behaviours, self-efficacy, perceived negative consequences associated with protective behaviours, reliance on sensory cue, and action planning. In addition, study participants who reported having a pre-existent respiratory condition and who were randomly allocated in the intervention group, also received specific additional messages targeting beliefs about efficacy and side effects of inhalers, and medication self-efficacy.

- Targeting message specificity:

Specificity refers to the extent to which a message provides a detailed description of the recommended behaviour. A meta-analysis of 18 studies (O'Keefe, 1997) found that messages providing health recommendations with a more specific description seem to be significantly more persuasive than generic recommendations (r=.10, k=18, N=11,105). Participants in the control group received the usual UK AQI message format containing less specific recommendations (e.g. advice for at risk individuals in case of high air pollution: 'Adults and children with lung problems, and adults with heart problems, should reduce strenuous physical exertion, particularly outdoors'). On the other hand, the intervention group received more specific recommendations ('Adults and children with lung problems, adults with heart problems, and older people, should reduce levels and length of physical activity outdoors. Where possible, change: travel route or exercise location (e.g. use our app to find less polluted roads or parks) or time (e.g. mornings or less polluted times)').

Control and intervention groups were compared in intended and actual behaviour change outcome measures. We predicted that the alternative format would be associated with higher behaviour change, compared to the usual format.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate, participants had to be members of the general public in the adult age range (>18 years), be fluent in English, working or living in Greater London, and being new or old users of a specific air quality alert smartphone application.

Exclusion Criteria:

* younger than 18 years
* not working or living in Greater London
* no longer users of the air quality alert smartphone application.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2017-07-23 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donatella D'Antoni, Principal Investigator — King's College London
Locations (1):
- King' College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] (WHO), W. H. O. (2014). Burden of disease from air pollution. Retrieved from http://www.who.int/phe/health_topics/outdoorair/databases/FINAL_HAP_AAP_BoD_24March2014.pdf?ua=1.
- [Background] D'Antoni D, Smith L, Auyeung V, Weinman J. Psychosocial and demographic predictors of adherence and non-adherence to health advice accompanying air quality warning systems: a systematic review. Environ Health. 2017 Sep 22;16(1):100. doi: 10.1186/s12940-017-0307-4. PMID 28938911
- [Background] Kelly FJ, Fussell JC. Air pollution and public health: emerging hazards and improved understanding of risk. Environ Geochem Health. 2015 Aug;37(4):631-49. doi: 10.1007/s10653-015-9720-1. Epub 2015 Jun 4. PMID 26040976
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Daniel J. O'Keefe (1997) Standpoint Explicitness and Persuasive Effect: A Meta-Analytic Review of the Effects of Varying Conclusion Articulation in Persuasive Messages, Argumentation and Advocacy, 34:1, 1-12, DOI: 10.1080/00028533.1997.11978023
- [Background] Samoli E, Atkinson RW, Analitis A, Fuller GW, Green DC, Mudway I, Anderson HR, Kelly FJ. Associations of short-term exposure to traffic-related air pollution with cardiovascular and respiratory hospital admissions in London, UK. Occup Environ Med. 2016 May;73(5):300-7. doi: 10.1136/oemed-2015-103136. Epub 2016 Feb 16. PMID 26884048

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants had to be members of the general public in the adult age range (> 18 years), be fluent in English, working or living in Greater London (as this is the geographical area that CityAir covers), and being new or existing users of the City Air smartphone application.
Pre-assignment Details: Of the 238 initially submitted questionnaires, 13 (5.5%) were incomplete, leaving a total of 225 complete initial questionnaires.
Period: Overall Study
Arm/Group | General Public/Usual Health Advice | General Public/Alternative Health Advice | At Risk Group/Usual Health Advice | At Risk Group/Alternative Health Advice
Started | 83 | 84 | 24 | 34
Final Questionnaire 4 Weeks Follow-up | 34 | 29 | 7 | 12
Completed | 34 | 29 | 7 | 12
Not Completed | 49 | 55 | 17 | 22
Not completed — Lost to Follow-up | 42 | 48 | 15 | 19
Not completed — Incomplete/unmatched questionnaire | 6 | 7 | 2 | 2
Not completed — Did not receive air alerts | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | General Public/Usual Health Advice | General Public/Alternative Health Advice | At Risk Group/Usual Health Advice | At Risk Group/Alternative Health Advice | Total
Number analyzed (Participants) | 34 | 29 | 7 | 12 | 82
Age, Customized [Count of Participants; unit: Participants]
  Age Range: 18-24 years | 0 | 2 | 0 | 0 | 2
  Age Range: 25-34 years | 12 | 12 | 1 | 5 | 30
  Age Range: 35-49 years | 17 | 11 | 1 | 3 | 32
  Age Range: 50+ years | 5 | 4 | 5 | 4 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 2 | 5 | 31
  Male | 21 | 18 | 5 | 7 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 31 | 27 | 6 | 10 | 74
  Ethnicity: Other | 3 | 2 | 1 | 2 | 8
Adoption of protective behaviour at baseline [Mean (Standard Deviation); unit: units on a scale] — Self-reported adoption of protective behaviours at baseline. Measures on a scale: from 1 Not at all to 9 all of the time (answers 'N/A, I am not aware of any forecast' were excluded from analyses). Participants were asked: 'In the past 4 weeks, how often have you taken action to reduce exposure to air pollution, in response to hearing or reading an air quality forecast?'
  units on a scale | 3.00 (0.45) | 2.38 (0.45) | 3.43 (1.42) | 2.83 (0.90) | 2.79 (0.30)

OUTCOME MEASURES:

1. Primary Outcome: Adoption of Protective Behaviour at 4 Weeks
Description: Differences between conditions in actual adoption of protective behaviours at 4 weeks. Outcome measures were collected via self-reports: The question was: 'In the past 4 weeks, how often have you taken action to reduce exposure to air pollution, in response to hearing or reading an air quality forecast?' Measures: from 1 'Not at all' to 9 'all of the time' (answers 'N/A, I am not aware of any forecast' were excluded from analyses).
Time Frame: Baseline and at 4 weeks
Population: ANCOVA (analysis of covariance) was performed for actual behaviour change at four weeks, adjusting for baseline data collected about one month earlier (target population and intervention/ control group were entered as fixed factors).
Measure: Mean (Standard Deviation); unit: units on a scale 1-9
Arm/Group | General Public/Usual Health Advice | General Public/Alternative Health Advice | At Risk Group/Usual Health Advice | At Risk Group/Alternative Health Advice
Number analyzed (Participants) | 34 | 29 | 7 | 12
units on a scale 1-9 | 3.67 (0.44) | 4.25 (0.48) | 4.29 (0.97) | 3.65 (0.74)
Statistical Analysis 1: Comparison: General Public/Usual Health Advice vs General Public/Alternative Health Advice vs At Risk Group/Usual Health Advice vs At Risk Group/Alternative Health Advice; We predicted that the groups receiving the alternative format of air quality notifications would report greater frequency of behaviour change at 4 weeks compared to the groups receiving the usual format; Test type: Other; p = .964, ANCOVA; ANCOVA, adjusted for baseline measures, tested for differences between intervention and control groups in preventative behaviours at 4 weeks

2. Secondary Outcome: Considered Making Permanent Changes
Description: Differences between conditions in planning the adoption of protective behaviours at 4 weeks. Outcome measures were collected via self-reports: The question was: 'In the past 4 weeks, have you considered making permanent changes to daily travel route or exercise location/time?' possible answers were 'yes' or 'no'. 'unsure' answers were treated as system missing.
Time Frame: at 4 weeks
Population: A Chi square test was performed to analyse whether there were significant differences in the proportion of respondents who had considered making permanent changes to their daily travel route, exercise location or exercise time between groups.
Measure: Count of Participants; unit: Participants
Arm/Group | General Public/Usual Health Advice | General Public/Alternative Health Advice | At Risk Group/Usual Health Advice | At Risk Group/Alternative Health Advice
Number analyzed (Participants) | 33 | 26 | 7 | 12
Participants
  yes | 10 | 14 | 3 | 7
  no | 23 | 12 | 4 | 5
Statistical Analysis 1: Comparison: General Public/Usual Health Advice vs General Public/Alternative Health Advice vs At Risk Group/Usual Health Advice vs At Risk Group/Alternative Health Advice; We predicted that more respondents in the intervention groups (i.e. receiving alternative health advice) would consider making permanent changes to their daily travel route, exercise location or exercise time compared to the control groups; Test type: Other; p = 0.043, Chi-squared; χ2(1)=4.11, V=0.229

3. Secondary Outcome: Actual Behaviour Change in Response to a Real Air Quality Alert
Description: Differences between conditions in self-reported actual behaviour change in response to receiving a real air quality alert. Behavioural outcomes were collected via a questionnaire asking participants to respond 'yes/no' to whether they had changed a series of behaviours in response to receiving the alert. In this case it was a 'moderate' alert
Time Frame: At 3 weeks
Population: Chi square tests were performed to analyse differences in proportion of self-reported actual behaviour change between groups, in relation to a real moderate air pollution episode. 'Unsure' answers in relation to actual behaviour change were treated as system missing and excluded from analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | General Public/Usual Health Advice | General Public/Alternative Health Advice | At Risk Group/Usual Health Advice | At Risk Group/Alternative Health Advice
Number analyzed (Participants) | 19 | 25 | 7 | 12
Participants
  Changed level/length of physical activity outdoors: number analyzed (Participants) | 19 | 25 | 6 | 12
  Changed level/length of physical activity outdoors: Yes | 3 | 2 | 2 | 5
  Changed level/length of physical activity outdoors: No | 16 | 23 | 4 | 7
  Changed travel route: number analyzed (Participants) | 19 | 25 | 7 | 11
  Changed travel route: Yes | 4 | 2 | 1 | 4
  Changed travel route: No | 15 | 23 | 6 | 7
  Changed travel time: number analyzed (Participants) | 19 | 25 | 7 | 11
  Changed travel time: Yes | 0 | 3 | 1 | 2
  Changed travel time: No | 19 | 22 | 6 | 9
  Changed exercise time: number analyzed (Participants) | 18 | 24 | 7 | 12
  Changed exercise time: Yes | 2 | 5 | 2 | 1
  Changed exercise time: No | 16 | 19 | 5 | 11
  Changed exercise location: number analyzed (Participants) | 17 | 24 | 7 | 11
  Changed exercise location: Yes | 2 | 6 | 2 | 1
  Changed exercise location: No | 15 | 18 | 5 | 10
Statistical Analysis 1: Comparison: General Public/Usual Health Advice vs General Public/Alternative Health Advice vs At Risk Group/Usual Health Advice vs At Risk Group/Alternative Health Advice; We predicted that the alternative health advice would lead to greater actual behaviour change compared to the usual format; Test type: Other; p > 0.05, Fisher Exact

4. Secondary Outcome: Intentions to Adhere to Health Advice Associated With a Hypothetical High Air Pollution Scenario
Description: Differences between conditions in intentions to adhere to the health advice received in association with a hypothetical high air pollution alert scenario. Intentions were measured by a self-report item: participants were asked to agree with a statement about their adherence intentions on 9-point scale, where 1=strongly disagree to 9=strongly agree.
Time Frame: Baseline and at 4 weeks
Population: ANCOVA (analysis of covariance) was performed for behavioural intentions in relation to the high air pollution hypothetical scenario at four weeks, adjusting for baseline data collected about one month earlier (target population and intervention/control group were entered as fixed factors).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | General Public/Usual Health Advice | General Public/Alternative Health Advice | At Risk Group/Usual Health Advice | At Risk Group/Alternative Health Advice
Number analyzed (Participants) | 34 | 29 | 7 | 12
score on a scale | 6.69 (0.23) | 6.26 (0.33) | 7.58 (0.28) | 6.93 (0.50)
Statistical Analysis 1: Comparison: General Public/Usual Health Advice vs General Public/Alternative Health Advice vs At Risk Group/Usual Health Advice vs At Risk Group/Alternative Health Advice; We predicted that the alternative format would lead to stronger intentions to adhere to recommendations associated with an hypothetical high air pollution episode compared to the usual format; Test type: Other; p > 0.05, ANCOVA; ANCOVA, adjusted for baseline intentions, tested for differences between groups in intentions in relation to an high-air-pollution scenario at 4 weeks

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | General Public/Usual Health Advice | General Public/Alternative Health Advice | At Risk Group/Usual Health Advice | At Risk Group/Alternative Health Advice
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT03552198/Prot_SAP_000.pdf